CLINICAL TRIAL: NCT06468800
Title: Feasibility and Added Value of the TRACMOTION Device for ESD
Acronym: TRACMOTION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Arjun D. Koch, MD, PhD, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL87167.078.24
Record Dates: First submitted 2024-06-11; First posted 2024-06-21 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Oesophageal Neoplasm
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ESD with TRACMOTION (Other): Patients already scheduled for ESD will undergo an ESD procedure with the aid of the TRACMOTION device.
  Interventions: Device: TRACMOTION

INTERVENTIONS:
Device: TRACMOTION — Patients already scheduled for ESD will undergo an ESD procedure with the aid of the Tracmotion device

SUMMARY:
A single center non-randomized prospective clinical study, to evaluate the feasibility and added value of the CE-certified Tracmotion device in patients scheduled consecutively for ESD in the upper and lower gastrointestinal tract.

After ESD, the endoscopists' opinion will be evaluated with a short questionnaire on experience with the Tracmotion device. The pathology report will be checked for radicality and microscopic damage of the removed lesion.

DETAILED DESCRIPTION:
Objective: The purpose of this study is to establish feasibility of the Tracmotion device for ESD and to define its added value during ESD in both upper and lower GI procedures, both in antegrade and in retroflex positions.

Study design: Single center prospective observational non-randomized clinical study.

Study population: A total of 20 consecutive cases scheduled for ESD will be included. Sample size calculation does not apply for this type of study. Patients already scheduled for ESD will undergo an ESD procedure as planned with the aid of the Tracmotion device. It is anticipated that the Tracmotion will provide superior traction and counter traction compared to off-label tools.

Intervention: Patients already scheduled for ESD will undergo an ESD procedure with the aid of the Tracmotion device.

Main study parameters/endpoints:

Feasibility: procedure time, dissection speed, lesional damage (tearing or grasping injury to the mucosa on macroscopy and pathological review) Added value: subjective evaluation of the Tracmotion device by the performing endoscopist (contentment of use of Tracmotion, difference in procedure time, stability of, control of and accessibility to the lesion).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for endoscopic submucosal dissection (upper and lower gastrointestinal tract);
* Lesion is accessible with a therapeutic endoscope;
* Written informed consent;
* Age ≥18 years.

Exclusion Criteria:

* Coagulopathy (not corrected prior to endoscopic submucosal dissection);
* Participating in a different experimental drug/device trial in the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Procedure time | During endoscopic submucosal dissection procedure
  Procedure time of the endoscopic submucosal dissection will be measured from start incision to end incision (in minutes)
Dissection speed | During endoscopic submucosal dissection procedure
  Dissection speed of ESD will be measured from start incision to end incision (square millimeter of dissected tissue per minute)
Lesional damage | During endoscopic submucosal dissection and during pathology review (on average 2 weeks after endoscopic submucosal dissection)
  Any tearing or grasping injury to the mucosa on macroscopy (yes vs. no) observed by the endoscopist and at pathological review (yes/no) observed by the pathologist expressed in percentages (%).
Subjective evaluation of the added value of the TRACMOTION device | Immediately after endoscopic submucosal dissection
  Directly after the endoscopic mucosal dissection the endoscopist will fill in a questionnaire using the Likert scale (1= worst experience possible, 5 = best experience possible) about their experience with the TRACMOTION device during ESD (overall contentment, difference of procedure time, stability of, control of and accessibility to the lesion that was resected)

SECONDARY OUTCOMES:
En-bloc rate | Determined Immediately after endoscopic submucosal dissection
  The incidence of en-bloc resections in percentages (%)
R0 rate | Determined during the pathology review (on average 2 weeks after endoscopic submucosal dissection)
  The incidence of R0 resections in percentages (%)
Complications after during and after endoscopic submucosal dissection | During endoscopic submucosal dissection procedure and 2 weeks after
  Complications will be measured during and after endoscopic submucosal dissection (bleeding yes/no, perforation yes/no) and will be expressed as percentages (%)

OTHER OUTCOMES:
Age | At baseline (after informed consent is signed)
  Age in years
Gender | At baseline (after informed consent is signed)
  Gender (male/female)
Tumor length | During endoscopic submucosal dissection, before incision starts
  Tumor length in millimeter (mm)
Tumor location | During endoscopic submucosal dissection, before incision starts
  Tumor location in centimeter (cm) measured from incisors
Tumor histology | After endoscopic submucosal dissection when the pathologist has reviewed the tissue (on average 2 weeks after endoscopic submucosal dissection)
  Tumor histology conform the pathology review
Prior treatment | At baseline (after informed consent is signed)
  Prior treatment of oesophageal neoplasms (such as chemotherapy, radiotherapy)
Use of symptomatic medication | 2 weeks after endoscopic submucosal dissection
  Use of symptomatic medication during 2 weeks after endoscopic submucosal dissection (analgesics, antiemetics, proton pump inhibitors)